CLINICAL TRIAL: NCT06180356
Title: Phase II Study to Assess the Efficacy of Niraparib Rechallenge After Surgery in Ovarian Cancer Patients With Oligometastatic Progression (The ANALLISA Study)
Brief Title: Niraparib Rechallenge After Surgery in Ovarian Cancer Patients With Oligometastatic Progression
Acronym: ANALLISA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDOPP557
Record Dates: First submitted 2023-12-01; First posted 2023-12-22 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer; Oligometastatic Disease; Serous Ovarian Tumor
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niraparib (Experimental)
  Interventions: Drug: Niraparib oral tablets

INTERVENTIONS:
Drug: Niraparib oral tablets — Niraparib 300 or 200 mg according to body weight or platelet count. Tablets will be taken orally, once daily, continuously (in 28-day cycles).

SUMMARY:
The ANALLISA study is a fast, proof-of-concept, phase II clinical trial which aims to assess the efficacy of niraparib rechallenge treatment after secondary cytoreductive surgery in ovarian cancer (OC) patients with oligometastatic progression (OMP) after first maintenance therapy with any PARP inhibitor. A total of 30 patients with OC and OMP will be enrolled and will receive treatment with niraparib 300 or 200 mg, according to body weight or platelet count. Patients will start treatment within 6 weeks after surgery and will receive it until progressive disease or treatment discontinuation. The main purpose of the study is to evaluate progression-free survival (PFS) of niraparib rechallenge in OC patients with OMP and no residual disease after secondary cytoreductive surgery.

DETAILED DESCRIPTION:
This is a single-arm phase II clinical trial which will enroll female patients aged ≥ 18 years with high grade serous or endometrioid ovarian cancer (OC) who have had an oligometastatic progression (OMP) during or after the first maintenance therapy with any poly adenosine diphosphate (ADP) ribose polymerase inhibitor (PARPi). OMP is defined as 1-5 metastatic lesions. Patients with symptomatic metastatic disease are not eligible.

A total of 30 patients with OC and OMP will be enrolled and will receive treatment with niraparib 300 or 200 mg, according to body weight or platelet count. Patients will start treatment within 6 weeks after surgery and will receive it until progressive disease or treatment discontinuation.

The main objective of the study is to evaluate progression-free survival (PFS) of niraparib rechallenge in OC patients with OMP and no residual disease after secondary cytoreductive surgery. Main secondary objectives are to assess the PFS according to biomarker status (BRCAm, BRCAwt, HRD and HRP), the PFS by CA 125, the second progression-free survival (PFS2), the time to start of first subsequent therapy or death (TFST) and the overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent form (ICF) prior to beginning specific protocol procedures.
2. Female patients ≥ 18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Patients must have a life expectancy ≥16 weeks.
5. Histologically confirmed high grade serous or endometrioid OC who have an OMP during or after the first maintenance therapy with any PARPi.
6. Oligometastatic progression defined as 1-5 lesions (according to European Society for Radiotherapy and Oncology [ESTRO] and American Society for Radiation Oncology [ASTRO] consensus).
7. Patients must have undergone secondary cytoreductive surgery with centrally confirmed no evidence of macroscopic residual tumor after surgery (complete resection).
8. Patients must have either normal or up to 2 x ULN CA 125 level.
9. Documented breast cancer gene 1/2 (BRCA1/2) status and homologous recombination (HR) status.
10. Patients who have received prior iPARP monotherapy or iPARP together with bevacizumab as maintenance treatment.
11. Patients should have had benefit of prior PARPi defined by exposure for ≥12 months (at least ≥ 18 months for patients who have a BRCA1/2 mutation) from initiation of PARPi maintenance until the date of OMP or have experienced a tumor progression after treatment completion. Tumor progression must have been confirmed by computed tomography (CT) and/or PET-CT scan.
12. If prior treatment was niraparib, no significant toxicity or need for treatment discontinuation was required.
13. Willingness to provide formalin fixed, paraffin embedded (FFPE) tumor tissue from primary, if available, and secondary surgeries and blood samples at screening, every 3 cycles (12 weeks), and at the end of treatment (EoT).
14. Able to take oral medications.
15. Patients must start treatment 3 to 6 weeks from surgery, once recovered from surgery.
16. Women of childbearing potential who engage in heterosexual intercourse must agree to use institution specified method(s) of contraception and must refrain from donating eggs in the time period specified in the study protocol. Women of childbearing potential must have a negative serum or a highly sensitive urine pregnancy test within 72 hours before study treatment initiation.
17. Patient has adequate bone marrow, liver, and renal function:

    * Hematological: White blood cell (WBC) count > 3.0 x 109/L, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100.0 x109/L, and hemoglobin ≥ 9.0 g/dL (≥ 5.6 mmol/L).
    * Hepatic: total bilirubin ≤ institutional upper limit of normal (ULN) (except for Gilbert's syndrome); alkaline phosphatase (ALP) ≤ 2.5 times ULN; aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 1.5 times ULN. 11).
    * Renal: serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
18. Patients must be accessible for treatment follow-up.

Exclusion Criteria:

1. Patients with symptomatic or systemic progressive disease not fulfilling OMP disease criteria.
2. Patients with residual disease after secondary cytoreductive surgery.
3. Patients with persistent toxicities (> Common Terminology Criteria for Adverse Events (CTCAE) grade 2) caused by previous cancer therapy.
4. Patients with central nervous system (CNS) metastases at baseline (post-secondary cytoreductive surgery).
5. Patients unable to swallow oral medication or with any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of niraparib, or put the study outcomes at undue risk.
6. Patients with clinically significant cardiovascular disease such as uncontrolled hypertension, uncontrolled or symptomatic arrythmias, congestive heart failure (CHF), or myocardial infarction within 6 months of screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association (NYHA) Functional Classification.
7. Patients treated with previous PARPi therapy who have any known, persistent (>4 weeks), ≥Grade 3 anemia, neutrophil count decrease or platelet count decrease.
8. Patients with known history of human immunodeficiency virus (HIV), or active hepatitis C Virus (HCV), or active hepatitis B Virus (HBV) infection, or any uncontrolled active systemic infection requiring intravenous antibiotics.
9. Patients with known hypersensitivity or allergy to prior niraparib treatment or any of the excipients of the product.
10. Patients who have received a transfusion of platelets or red blood cells, colony-stimulating factors or have any other laboratory abnormality within 2 weeks prior niraparib treatment that might confound or interfere with the study result.
11. Patients must not be simultaneously enrolled in any clinical trial of niraparib or any other investigational therapy.
12. Patients who are pregnant or breastfeeding or expecting to conceive children within the projected duration of the study treatment.
13. Patients with myelodysplastic syndrome (MSD)/Acute myeloid leukemia (AML), with history of MSD/AML or with features suggestive of MDS/AML.
14. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
15. Other malignancy unless curatively treated with no evidence of disease ≥ 5 years prior to study enrollment. Note: Patients with adequately non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS) and stage 1 low grade endometrial carcinoma are not excluded.
16. Vaccination with any live virus vaccine within 28 days prior study treatment initiation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Baseline up to 7 months
  PFS is defined as the period of time from niraparib treatment initiation until the subsequent disease progression or death, whichever occurs first, as determined locally by the investigator through the use of Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v.1.1)

SECONDARY OUTCOMES:
Progression free-survival according to biomarker status (BRCAm, BRCAwt, HRD and HRP) | Baseline up to 7 months
  PFS by biomarker status is defined as the period of time from niraparib treatment initiation until the subsequent disease progression or death, whichever occurs first, as determined locally by the investigator through the use of RECIST v.1.1, in patients' subgroups
Progression free-survival by CA 125 | Baseline up to 7 months
  PFS by CA 125 is defined as the time from treatment initiation until disease progression or death, whichever occurs first, as determined locally by the investigator using Gynecologic Cancer Intergroup (GCIC) criteria for CA 125 biomarker
Second progression-free survival (PFS2) | Baseline up to 7 months
  PFS2 is defined as the time from treatment initiation to the earliest progression event after that used for the primary variable PFS, or date of death as determined locally by the investigator using RECIST v.1.1
Time to start of first subsequent therapy or death (TFST) | Baseline up to 7 months
  TFST is defined as the time from the date of treatment initiation to the earliest date of anti-cancer therapy start date following study treatment discontinuation, or death
Overall survival (OS) | Baseline up to 7 months
  OS is defined as the period from treatment initiation to death from any cause, as determined locally by the investigator
Incidence of Adverse Events, Serious Adverse Events and Suspected Unexpected Serious Adverse Reactions | Baseline up to 7 months
  Number of Adverse Events (AEs), Serious Adverse Events (SAEs), and Suspected Unexpected Serious Adverse Reactions (SUSARs) according to the National Cancer Institute (NCI) CTCAE Version 5.0 (v.5.0) (Safety and Tolerability)

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Cortés Salgado, Principal Investigator — Hospital Universitario Ramón y Cajal, IRYCIS, Madrid (Spain)
Locations (14):
- Spain (14):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital de Cruces, Barakaldo
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Institut Català d' Oncologia Girona (ICO), Girona
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Central de Asturias (HUCA), Oviedo
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari Sant Joan de Reus, Tarragona
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No